CLINICAL TRIAL: NCT06349512
Title: 68Ga-FAPI-46 PET/CT for Predicting Histological Response to Neoadjuvant Chemo-immunotherapy in Triple-negative Breast Cancer
Brief Title: 68Ga-FAPI-46 PET/CT for Predicting Histological Response in Triple-negative Breast Cancer (FAP-IT)
Acronym: FAP-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2022-07; 2023-507860-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective multicenter study evaluating the prediction of histological response after neoadjuvant pembrolizumab in combination with chemotherapy by pre-treatment 68Ga-FAPI-46 PET/CT imaging in patients with early-stage high-risk TNBC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triple Negative Breast Cancer (Experimental): Patients with early-stage high-risk Triple Negative Breast Cancer
  Interventions: Procedure: 68Ga-FAPI-46 PET/CT imaging

INTERVENTIONS:
Procedure: 68Ga-FAPI-46 PET/CT imaging — The 68Ga-FAPI-46 PET/CT scan will be performed for each patient pre-therapy and on the same machine as the 18F-FDG PET/CT scan and within 14 days before the start of treatment.

SUMMARY:
Prospective multicenter study evaluating the prediction of histological response after neoadjuvant pembrolizumab in combination with chemotherapy by pre-treatment 68Ga-FAPI-46 PET/CT imaging in patients with early-stage high-risk TNBC.

DETAILED DESCRIPTION:
Prospective multicenter study evaluating the prediction of histological response of pembrolizumab in combination with neoadjuvant chemotherapy by pre-treatment 68Ga-FAPI-46 PET/CT imaging in patients with early-stage high-risk TNBC.

Patients will receive the newly established standard of care of neoadjuvant pembrolizumab 200 mg Q3W given with 4 cycles of paclitaxel + carboplatin, then with 4 cycles of doxorubicin or epirubicin + cyclophosphamide. After definitive surgery, patients will receive adjuvant pembrolizumab for 9 cycles or until recurrence or unacceptable toxicity.

The 68Ga-FAPI-46 PET/CT scan will be performed for each patient pre-therapy and on the same machine as the 18F-FDG PET/CT scan and within 14 days before the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female with age ≥ 18 years,
2. Patients with previously untreated, non-metastatic, centrally confirmed TNBC for whom a neoadjuvant treatment with chemotherapy + pembrolizumab is the recommended option as standard of care,
3. Patients with measurable targets according to RECIST/PERCIST criteria,
4. Patients without distant metastasis based on staging 18F-FDG PET/CT,
5. Patients with tumor tissue available,
6. Patients who provided a signed written informed consent,
7. Patient ability to comply with protocol requirements,
8. Patients covered by a health insurance system.

Exclusion Criteria:

1. Pregnant and lactating women,
2. Patients with prior anti-PD(L)1 immunotherapy,
3. Patients with any contra-indication to chemo-immunotherapy standard of care therapy, per investigator assessment,
4. Patients with altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient informed consent,
5. Patients who have difficulty undergoing trial procedures for geographic, social or psychological reasons,
6. Person deprived of liberty or under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female are included
Enrollment: 60 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2032-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve | 6 months
  To measure the performance of 68Ga-FAPI-46 PET/CT imaging to predict complete histological response after neoadjuvant chemotherapy plus Pembrolizumab, in terms of Area under the ROC curve (AUC of the ROC curve).

SECONDARY OUTCOMES:
Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT performances | Baseline
  Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT performances by detecting metastases
Evaluation of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT performances | Baseline
  Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT performances by evaluating the tumor burden (TFTV : total FAP expression tumor volume and TMTV : total metabolic tumor volume).
Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT predictive performances | Day 168
  Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT predictive performances, separately and combined at the end of neoadjuvant treatment cycles.
Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT pronostic performances | 5 years
  Comparison of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT pronostic performances, separately and combined at the end of the follow-up
Evaluation of predictive model performance combining 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT | Baseline
  Evaluation of predictive model performance combining 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT imaging data, using sensitivity, specificity, positive and negative predictive values and area under the ROC curve (AUC of the ROC curve)

CONTACTS AND LOCATIONS:
Overall Officials: Romain-David SEBAN, Principal Investigator — Institut Curie
Locations (6):
- France (6):
  - Hôpital Privé d'Antony, Antony
  - Institut Curie -site Paris, Paris
  - GH Diaconesses Croix Saint-Simon, Paris
  - Institut Curie -site St Cloud, Saint-Cloud
  - HIA Begin, Saint-Mandé
  - Hôpital FOCH, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified data sets with interested researchers, educators or clinicians. Materials generated under the project will be disseminated in accrodance with Institut Curie policies.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific reserach, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).